CLINICAL TRIAL: NCT04913857
Title: New Wine in Old Bottle: the Effects of SUDOKU Mind Activation and Revitalizing Training (SMART) Program on Cognitive Function Among People With Mild Cognitive Impairment
Brief Title: Effects of SUDOKU Mind Activation & Revitalizing Training on Cognitive Function in People With Mild Cognitive Impairment
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMART
Record Dates: First submitted 2021-04-16; First posted 2021-06-04 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: To implement a SMART Program to promote cognitive health among patients with MCI, and the use of active mind strategy in preventing dementia among the older adults
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24-week SUDOKU Training Programme (Experimental): The SUDOKU training program include a 12-week face-to-face training session and a 12-week facilitated self-practice. The 12-week (60-minute sessions) training program will be evenly divided into 3 modules of increasing difficulty for the suboptimal cognitive function of the participants with MCI. As the use of T-code in solving the SUDOKU allows communicating the way a number is assigned to a box, participants are grouped into a small team of 3, so that they will work together during the tutorial practice.
  Facilitated self-practice will last for another 12 weeks immediately after the group training session. The instructor will give them a workbook with 12 SUDOKU puzzles of increasing level of difficulty for completion. The instructor will encourage and facilitate their accomplishment by giving them guidance on the taught method through regular phone call. Solutions of the assigned puzzle and the T-code will be provided in the following week.
  Interventions: Behavioral: 24-week SUDOKU Training Programme
- wait-list (Active Comparator): wait-list comparison group will receive the same program upon completion of the 6-month posttest evaluation on study outcomes
  Interventions: Other: Control Arm (wait-list)

INTERVENTIONS:
Behavioral: 24-week SUDOKU Training Programme — 12-week face-to-face training session and a 12-week facilitated self-practice
  Other Names: SMART
  Arms: 24-week SUDOKU Training Programme
Other: Control Arm (wait-list) — wait-list comparison group will receive the same program upon completion of the 6-month posttest evaluation on study outcomes
  Arms: wait-list

SUMMARY:
This study aims to implement a SUDOKU Mind Activation and Revitalization Training (SMART) Program to promote cognitive health among patients with mild cognitive impairment (MCI), and the use of active mind strategy in preventing dementia among the older adults. The SMART Program consists of two components including, a community empowerment-educational campaign on active mind strategies for older adults, and a 24-week SUDOKU Training Programme for people with MCI.

DETAILED DESCRIPTION:
This study aims to implement a SMART Program to promote cognitive health among patients with MCI, and the use of active mind strategy in preventing dementia among the older adults. The SMART Program consists of two components including, a community empowerment-educational campaign on active mind strategies for older adults, and a 24-week SUDOKU Training Programme for people with MCI.

The community empowerment-educational campaign will be conducted in the elderly care centres of the two collaborating non-governmental organizations, with the purpose of increasing the awareness of people aged 55 or above on the importance of maintaining an active mind and preventing age-related cognitive decline and dementia. The campaign will include cognitive screening, poster exhibition, booth exhibition and individual counselling.

The SUDOKU training program include a 12-week face-to-face training session and a 12-week facilitated self-practice. The face-to-face sessions aim at developing the skills of the participants in solving the SUDOKU using the T-code. The 12-week training program will be evenly divided into three modules of increasing difficulty, with consideration given to the suboptimal cognitive function of the participants with MCI. These modules are developed by the Co-investigator who has rich prior experience in teaching older adults on SUDOKU puzzle.

ELIGIBILITY:
Inclusion Criteria:

* People with MCI as defined by a score of 19-26 out of the 30 on the Montreal Cognitive Assessment in the general public and aged 55 or above.

Exclusion Criteria:

* Persons with dementia and communication problems will be excluded.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cantonese version of the Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | Baseline
  To evaluate various domains of cognition
Cantonese version of the Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | 12-week
  To evaluate various domains of cognition
Cantonese version of the Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | 24-week
  To evaluate various domains of cognition
The digit span-forward and backward test | Baseline
  To measure attention and working memory
The digit span-forward and backward test | 12-week
  To measure attention and working memory
The digit span-forward and backward test | 24-week
  To measure attention and working memory
The list learning delayed recall test | Baseline
  To measure episodic memory
The list learning delayed recall test | 12-week
  To measure episodic memory
The list learning delayed recall test | 24-week
  To measure episodic memory
Trail-Making Test Part A and B | Baseline
  To measure complex attention, executive function and task switching
Trail-Making Test Part A and B | 12-week
  To measure complex attention, executive function and task switching
Trail-Making Test Part A and B | 24-week
  To measure complex attention, executive function and task switching

SECONDARY OUTCOMES:
Memory Inventory for Chinese | Baseline
  To evaluate the subjective memory impairment
Memory Inventory for Chinese | 12-week
  To evaluate the subjective memory impairment
Memory Inventory for Chinese | 24-week
  To evaluate the subjective memory impairment
The 36-item Chinese version of the Short Form 36 (SF-36) | Baseline
  To measure Health-related quality of life in the participants
The 36-item Chinese version of the Short Form 36 (SF-36) | 24-week
  To measure Health-related quality of life in the participants

OTHER OUTCOMES:
13-item satisfaction survey - for SMART Program | 12-week
  To evaluate the participant's satisfaction towards the Sudoku program including acceptability, applicability to promote brain health and psychosocial health, accessibility and level of support
10-item satisfaction survey - for community empowerment-educational campaign | 10-month
  To evaluate the participant's satisfaction towards this service component

CONTACTS AND LOCATIONS:
Overall Officials: Doris, Sau Fung YU, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine and Geriatrics, United Christian Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Only study investigators and research assistants involved in the study will have access to the data.

REFERENCES:
- [Background] Wu YT, Lee HY, Norton S, Chen C, Chen H, He C, Fleming J, Matthews FE, Brayne C. Prevalence studies of dementia in mainland china, Hong Kong and taiwan: a systematic review and meta-analysis. PLoS One. 2013 Jun 11;8(6):e66252. doi: 10.1371/journal.pone.0066252. Print 2013. PMID 23776645
- [Background] Lam LC, Tam CW, Lui VW, Chan WC, Chan SS, Wong S, Wong A, Tham MK, Ho KS, Chan WM, Chiu HF. Prevalence of very mild and mild dementia in community-dwelling older Chinese people in Hong Kong. Int Psychogeriatr. 2008 Feb;20(1):135-48. doi: 10.1017/S1041610207006199. Epub 2007 Sep 25. PMID 17892609
- [Background] Ding D, Zhao Q, Guo Q, Liang X, Luo J, Yu L, Zheng L, Hong Z; Shanghai Aging Study (SAS). Progression and predictors of mild cognitive impairment in Chinese elderly: A prospective follow-up in the Shanghai Aging Study. Alzheimers Dement (Amst). 2016 Apr 9;4:28-36. doi: 10.1016/j.dadm.2016.03.004. eCollection 2016. PMID 27489876
- [Background] Wirth M, Haase CM, Villeneuve S, Vogel J, Jagust WJ. Neuroprotective pathways: lifestyle activity, brain pathology, and cognition in cognitively normal older adults. Neurobiol Aging. 2014 Aug;35(8):1873-82. doi: 10.1016/j.neurobiolaging.2014.02.015. Epub 2014 Feb 20. PMID 24656834
- [Background] Reuter-Lorenz PA, Park DC. How does it STAC up? Revisiting the scaffolding theory of aging and cognition. Neuropsychol Rev. 2014 Sep;24(3):355-70. doi: 10.1007/s11065-014-9270-9. Epub 2014 Aug 21. PMID 25143069
- [Background] Sherman DS, Mauser J, Nuno M, Sherzai D. The Efficacy of Cognitive Intervention in Mild Cognitive Impairment (MCI): a Meta-Analysis of Outcomes on Neuropsychological Measures. Neuropsychol Rev. 2017 Dec;27(4):440-484. doi: 10.1007/s11065-017-9363-3. Epub 2017 Dec 27. PMID 29282641
- [Background] Tardif S, Simard M. Cognitive stimulation programs in healthy elderly: a review. Int J Alzheimers Dis. 2011;2011:378934. doi: 10.4061/2011/378934. Epub 2011 Aug 15. PMID 21876829
- [Background] Brooker H, Wesnes KA, Ballard C, Hampshire A, Aarsland D, Khan Z, Stenton R, McCambridge L, Corbett A. An online investigation of the relationship between the frequency of word puzzle use and cognitive function in a large sample of older adults. Int J Geriatr Psychiatry. 2019 Jul;34(7):921-931. doi: 10.1002/gps.5033. Epub 2019 May 16. PMID 30443984
- [Background] Schultz SA, Larson J, Oh J, Koscik R, Dowling MN, Gallagher CL, Carlsson CM, Rowley HA, Bendlin BB, Asthana S, Hermann BP, Johnson SC, Sager M, LaRue A, Okonkwo OC. Participation in cognitively-stimulating activities is associated with brain structure and cognitive function in preclinical Alzheimer's disease. Brain Imaging Behav. 2015 Dec;9(4):729-36. doi: 10.1007/s11682-014-9329-5. PMID 25358750
- [Background] Pillai JA, Hall CB, Dickson DW, Buschke H, Lipton RB, Verghese J. Association of crossword puzzle participation with memory decline in persons who develop dementia. J Int Neuropsychol Soc. 2011 Nov;17(6):1006-13. doi: 10.1017/S1355617711001111. PMID 22040899
- [Background] Ferreira N, Owen A, Mohan A, Corbett A, Ballard C. Associations between cognitively stimulating leisure activities, cognitive function and age-related cognitive decline. Int J Geriatr Psychiatry. 2015 Apr;30(4):422-30. doi: 10.1002/gps.4155. Epub 2014 Jul 3. PMID 24989949
- [Background] Chu LW, Chiu KC, Hui SL, Yu GK, Tsui WJ, Lee PW. The reliability and validity of the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) among the elderly Chinese in Hong Kong. Ann Acad Med Singap. 2000 Jul;29(4):474-85. PMID 11056778
- [Background] Lui VW, Lam LC, Chiu HF. Validation of a memory inventory for the assessment of awareness of memory deficits in Alzheimer's disease in Chinese elderly. Int J Geriatr Psychiatry. 2006 Oct;21(10):917-23. doi: 10.1002/gps.1580. PMID 16927409
- [Background] Lam CL, Gandek B, Ren XS, Chan MS. Tests of scaling assumptions and construct validity of the Chinese (HK) version of the SF-36 Health Survey. J Clin Epidemiol. 1998 Nov;51(11):1139-47. doi: 10.1016/s0895-4356(98)00105-x. PMID 9817131
- [Background] Rabiee F. Focus-group interview and data analysis. Proc Nutr Soc. 2004 Nov;63(4):655-60. doi: 10.1079/pns2004399. PMID 15831139
- See also: Global Council on Brain Health. "Engaging your brain: GCBH recommendations on cognitively stimulating activities." — http://www.GlobalCouncilOnBrainHealth.org
- See also: Lam J. Numbers add up for scores of seniors in Sudoku competition. — http://www.thestandard.com.hk

DOCUMENTS (1):
  • Informed Consent Form (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT04913857/ICF_000.pdf